CLINICAL TRIAL: NCT01299259
Title: Improving Primary Care Follow-up for Adolescents With PID: A Randomized Controlled Trial Using Text Message Reminders
Brief Title: Improving Primary Care Follow-up for Patients With Pelvic Inflammatory Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 10-007744
Record Dates: First submitted 2010-11-30; First posted 2011-02-18 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Pelvic Inflammatory Disease
Keywords: Text message reminders; Pelvic inflammatory disease; PID; Primary care follow-up; Emergency department care; Discharge instructions
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Text Message Reminders (Experimental): Subjects randomized to the the intervention group will receive a total of 4 text messages on days 2 through 5 to remind them to schedule and attend a PCP follow-up appointment
  Interventions: Behavioral: Text Message Reminders
- Control Group (No Intervention): The control group will not receive any additional reminders to follow-up with PCP.

INTERVENTIONS:
Behavioral: Text Message Reminders — Patients in the intervention group will receive text messages on their cell phones following discharge from the emergency department reminding them to make an appointment with their primary care provider. Text messages will be sent daily for 4 days after discharge from the ED.
  Arms: Text Message Reminders

SUMMARY:
The investigators hypothesize that text message reminders to girls diagnosed with pelvic inflammatory disease (PID) in the emergency department (ED) will improve follow-up to their primary care provider (PCP) after being discharged from the ED.

DETAILED DESCRIPTION:
The Centers for Disease Control (CDC) recommends that patients diagnosed with pelvic inflammatory disease (PID) receive follow-up care within 72 hours of diagnosis. However, recent studies show that the majority of teenage girls diagnosed with PID do not receive this follow-up care within 72 hours. We hypothesize that text message reminders to girls diagnosed with PID in the emergency department (ED) will improve follow-up to their primary care provider (PCP) after being discharged from the ED.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 15 years and older
* New diagnosis of PID, as defined by the 2006 CDC minimum criteria for diagnosis of PID, on current ED encounter
* Determined by attending physician to be appropriate for outpatient treatment

Exclusion Criteria:

* Patient does not have a cell phone that is capable of receiving text messages
* Developmental disability
* Non-English speaking
* Pregnancy
* Patient who was enrolled in this study on a prior ED visit

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
PCP follow-up rates will be used to evaluate the efficacy of text message reminders. | PCP follow-up rates will be assessed 7-14 days after discharge from the ED.

SECONDARY OUTCOMES:
Number of adolescents who accept text message reminders as an measure of feasibility and acceptability. | 7-14 days after discharge from the ED
  The acceptability among adolescents of using text message reminders after ED discharge in adolescents treated in a pediatric ED.
Number of adolescents satisfied with ED care between the control group and intervention group as a measure of patient satisfaction. | 7-14 days after ED discharge
  Patient satisfaction of ED care when receiving text message reminders.
Type of participant characteristics associated with PCP follow-up as a measure of behavior change, compliance and rate of follow-up care | 7-14 days after ED discharge
  Patient characteristics associated with PCP follow-up
Barriers to PCP follow-up from an ED visit to measure use of text message technology and rate of change in follow-up care between groups | 7-14 days after ED visit
  Types of barriers encountered to PCP follow-up from an ED visit for PID care to measure rate of change in follow-up care between groups

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Mollen, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia; Frances Balamuth, MD, PhD, Study Director — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention; Workowski KA, Berman SM. Sexually transmitted diseases treatment guidelines, 2006. MMWR Recomm Rep. 2006 Aug 4;55(RR-11):1-94. PMID 16888612
- [Background] Trent M, Ellen JM, Walker A. Pelvic inflammatory disease in adolescents: care delivery in pediatric ambulatory settings. Pediatr Emerg Care. 2005 Jul;21(7):431-6. doi: 10.1097/01.pec.0000169432.14067.eb. PMID 16027575
- [Background] Trent M, Judy SL, Ellen JM, Walker A. Use of an institutional intervention to improve quality of care for adolescents treated in pediatric ambulatory settings for pelvic inflammatory disease. J Adolesc Health. 2006 Jul;39(1):50-6. doi: 10.1016/j.jadohealth.2005.08.008. PMID 16781961
- [Background] Engel KG, Heisler M, Smith DM, Robinson CH, Forman JH, Ubel PA. Patient comprehension of emergency department care and instructions: are patients aware of when they do not understand? Ann Emerg Med. 2009 Apr;53(4):454-461.e15. doi: 10.1016/j.annemergmed.2008.05.016. Epub 2008 Jul 10. PMID 18619710
- [Background] Armstrong AW, Watson AJ, Makredes M, Frangos JE, Kimball AB, Kvedar JC. Text-message reminders to improve sunscreen use: a randomized, controlled trial using electronic monitoring. Arch Dermatol. 2009 Nov;145(11):1230-6. doi: 10.1001/archdermatol.2009.269. PMID 19917951
- [Background] Franklin VL, Greene A, Waller A, Greene SA, Pagliari C. Patients' engagement with "Sweet Talk" - a text messaging support system for young people with diabetes. J Med Internet Res. 2008 Jun 30;10(2):e20. doi: 10.2196/jmir.962. PMID 18653444
- [Background] Miloh T, Annunziato R, Arnon R, Warshaw J, Parkar S, Suchy FJ, Iyer K, Kerkar N. Improved adherence and outcomes for pediatric liver transplant recipients by using text messaging. Pediatrics. 2009 Nov;124(5):e844-50. doi: 10.1542/peds.2009-0415. Epub 2009 Oct 12. PMID 19822583
- [Background] Riley W, Obermayer J, Jean-Mary J. Internet and mobile phone text messaging intervention for college smokers. J Am Coll Health. 2008 Sep-Oct;57(2):245-8. doi: 10.3200/JACH.57.2.245-248. PMID 18809542
- [Derived] Wolff M, Balamuth F, Sampayo E, Mollen C. Improving Adolescent Pelvic Inflammatory Disease Follow-up From the Emergency Department: Randomized Controlled Trial With Text Messages. Ann Emerg Med. 2016 May;67(5):602-609.e3. doi: 10.1016/j.annemergmed.2015.10.022. Epub 2015 Dec 11. PMID 26686262